CLINICAL TRIAL: NCT01600131
Title: Utilizing the RESCUE Stroke Caregiver Website to Enhance Discharge Planning
Brief Title: RESCUE Stroke Caregiver Website to Enhance Discharge Planning
Acronym: RESCUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IIR 11-343
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Results first posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2022-04

CONDITIONS: Depression; Quality of Life; Self Efficacy; Recovery of Function; Stress; Positive Aspects of Caregiving
MeSH Terms: conditions — Depression | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Caregiver education and support (Experimental): problem-solving intervention for stroke caregivers that can be delivered shortly after the Veteran's in-patient stays followed by online, in-home sessions. The investigators will modify the traditional, problem-solving intervention by adding web-based training using interactive modules, factsheets, and tools on the investigators' previously developed and nationally available RESCUE Caregiver website (www.cidrr8.research.va.gov/rescue). The investigators will also provide on-line, skills training and application of the problem-solving approach via the RESCUE messaging center.
  Interventions: Behavioral: Caregiver problem-solving
- Standard Care (Other): Caregivers receiving standard of care
  Interventions: Other: Standard Care

INTERVENTIONS:
Behavioral: Caregiver problem-solving — This is a problem-solving intervention for stroke caregivers that can be delivered shortly after the Veteran's in-patient stays followed by online, in-home sessions. The investigators will modify the traditional, problem-solving intervention by adding web-based training using interactive modules, factsheets, and tools on the investigators' previously developed and nationally available RESCUE Caregiver website (www.ciddr8.research.va.gov/rescue). The investigators will also provide on-line, skills training and application of the problem-solving approach via the RESCUE messaging center.
  Arms: Caregiver education and support
Other: Standard Care — No intervention or treatment will be provided. The investigators will closely monitor the usual care that is provided to caregivers.
  Arms: Standard Care

SUMMARY:
Aims and Intervention:

The long-term goal is to implement stroke caregiver programs that involve low-cost interventions that are sustainable in routine clinical practice. The immediate objective is to test, using a randomized controlled trial, a problem-solving intervention for stroke caregivers that can be delivered during the transitional care period (e.g., time which Veteran is discharged to home) followed by online, in-home sessions. The investigators will modify the traditional, problem-solving intervention by adding web-based training using interactive modules, factsheets, and tools on previously developed and nationally available RESCUE Caregiver website (www.cidrr8.research.va.gov/rescue). The investigators will also provide on-line, skills training and application of the problem-solving approach via the RESCUE messaging center. The immediate, primary aim (#1) is to test the effect of the intervention on stroke caregivers' depressive symptoms at 11 and 19 weeks after baseline data collection. Aim #2 is to test the effect of the intervention on stroke caregivers' burden, positive aspects of caregiving, self-efficacy, health-related quality of life (HRQOL), and satisfaction with care at 11 and 19 weeks after baseline data collection. Aim #3 is to test the effect of the intervention on Veterans' outcomes: functional abilities and healthcare utilization (i.e., unintended hospital bed days of care, number of emergency room visits, number of unscheduled clinic visits) at 11 and 19 weeks after baseline data collection. Aim #4 is to determine the budgetary impact for implementing the intervention. Aim #5 is to determine the facilitators, barriers and best practices for implementing the intervention.

Design and Methods:

The investigators will conduct a two-group randomized controlled trial. The investigators will enroll 240 stroke caregivers at 8 study sites (North Florida/South Georgia Veterans Healthcare System, Miami VA Healthcare System, James A. Haley Veterans Hospital in Tampa, Michael E. Debakey VAMC in Houston, Hunter Holmes McGuire VAMC in Richmond, Central Arkansas Veterans Healthcare System, VA Tennessee Valley Healthcare System, and the VA Boston Healthcare System). Eligible caregivers will be interviewed, complete baseline measures, and then be randomized to two groups: 1) intervention group, or 2) standard care. A team member will telephone caregivers at 11 weeks and 19 weeks after baseline data collection to answer questions on instruments with established reliability and validity. Qualitative interviews will be conducted with selected caregivers to obtain in-depth perceptions of the value, facilitators, and barriers of the intervention.

Impact:

This is the first known study to test a transition-to-home intervention combined with technology to improve the quality of caregiving and the recovery of Veterans.

DETAILED DESCRIPTION:
Background:

Caregiver depression is common following a family member's stroke and is a major contributor of survivor's hospital readmission and institutionalization. Researchers have consistently found that interventions to help caregivers resolve problems are effective in reducing depressive symptoms. However, these problem-solving interventions have been underused in practice because they involve multiple, in-person or telephone sessions and require large amounts of staff time to implement. To overcome these barriers, the long-term goal is to implement stroke caregiver programs that involve low-cost interventions that are sustainable in routine clinical practice. The immediate objective is to test, using a randomized controlled trial, a problem-solving intervention for stroke caregivers that can be delivered shortly after the Veterans' in-patient stays followed by online, in-home sessions. The investigators will modify the traditional, problem-solving intervention by adding web-based training using interactive modules, factsheets, and tools on previously developed and nationally available RESCUE Caregiver website (www.cidrr8.research.va.gov/rescue). The investigators will also provide on-line, skills training and application of the problem-solving approach via the RESCUE messaging center, a secure site behind the VA firewall. This work builds on the team's extensive experience in stroke caregiver education.

The immediate, primary aim (#1) is to test the effect of the intervention on stroke caregivers' depressive symptoms at 11 and 19 weeks after baseline data collection. Primary Hypothesis: Stroke caregivers who receive the intervention will have less depressive symptoms at 11 and 19 weeks after baseline data collection compared to stroke caregivers who receive standard care. The investigators propose four secondary aims. Aim #2 is to test the effect of the intervention on stroke caregivers' burden, positive aspects of caregiving, self-efficacy, health-related quality of life (HRQOL), and satisfaction with care at 11 and 19 weeks after baseline data collection. Aim #3 is to test the effect of the intervention on Veterans' outcomes: functional abilities and healthcare utilization (i.e., unintended hospital bed days of care, number of emergency room visits, number of unscheduled clinic visits) at 11 and 19 weeks after baseline data collection. Aim #4 is to determine the budgetary impact for implementing the intervention. Aim #5 is to determine the facilitators, barriers and best practices for implementing the intervention.

Methods:

The investigators will conduct a two-group randomized controlled trial with repeated measures and use mixed methods to determine caregivers' perceptions of the intervention. The investigators will enroll 240 stroke caregivers at 8 study sites (North Florida/South Georgia Veterans Healthcare System, Miami VA Healthcare System, James A. Haley Veterans Hospital in Tampa, Michael E. Debakey VAMC in Houston, Hunter Holmes McGuire VAMC in Richmond, Central Arkansas Veterans Healthcare System, VA Tennessee Valley Healthcare System, and the VA Boston Healthcare System). Eligible caregivers will be interviewed, complete baseline measures, and then be randomized to two groups: 1) intervention group, or 2) standard care. A study team member will telephone caregivers at 11 weeks and 19 weeks after baseline data collection to answer questions on instruments with established reliability and validity. The team member will review the Veterans' VA Computerized Patient Record System health record to obtain information on the Veterans' healthcare utilization. The investigators will determine the budgetary impact of the intervention by examining the cost data in the VA Managerial Cost Accounting System (MCAS) (formerly DSS) National Data Extracts and Non-VA Medical Care files. Qualitative interviews will be conducted with selected caregivers to obtain in-depth perceptions of the value, facilitators, and barriers of the intervention. Throughout all phases of the project, the investigators will collaborate with VA (Offices of Nursing Service and Office of Geriatrics and Extended Care.

Impact:

This is the first known study to test transition-to-home intervention combined with technology to improve the quality of caregiving and the recovery of Veterans. Other outcomes will be a state-of-the-art website and an evidence-based model (in-patient, discharge planning and online, training and caregiver-provider messaging) that can be transportable to other disease models

ELIGIBILITY:
Inclusion Criteria:

All caregivers of Veterans with a primary diagnosis of stroke are eligible for participation if they meet the following criteria:

* are the primary caregiver and provide the majority of care for a Veteran who has a primary diagnosis of stroke (ICD9 codes for stroke: 430-438) and who has at least one activity of daily living (ADL) deficits or a new or worsening cognitive or physical functioning problem,
* have Internet and email access and ability,
* are reachable by cell or home phone,
* read English at the sixth grade reading level or better,
* score 1 or greater on the Perceived Stress Scale
* Veteran has been discharged to home within the preceding four months or plans to be ultimately discharged to home
* are agreeable to be randomized to the intervention or standard care group

Exclusion Criteria:

Caregivers who fail to meet one or more of the inclusion criteria and whose Veterans

* are terminally ill
* have a life expectancy of less than 6 months
* are a prisoner, or
* are professional caregivers who had no preexisting relationship to the Veteran
* are enrolled or have completed similar caregiving interventions (at PI discretion)

Life expectancy and service use will be determined by reviewing the CPRS records and conferring with the in-patient staff and with the investigators' clinical team members (MDs, RNs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2015-06-22 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Constance R. Uphold, PhD MS BS, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (3):
- United States (3):
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Graf R, LeLaurin J, Schmitzberger M, Freytes IM, Orozco T, Dang S, Uphold CR. The stroke caregiving trajectory in relation to caregiver depressive symptoms, burden, and intervention outcomes. Top Stroke Rehabil. 2017 Oct;24(7):488-495. doi: 10.1080/10749357.2017.1338371. Epub 2017 Jun 15. PMID 28618848
- [Result] LeLaurin J, Schmitzberger M, Eliazar-Macke N, Freytes IM, Dang S, Uphold C. A commentary on methodological issues in stroke caregiver research: lessons learned from three RESCUE intervention studies. Top Stroke Rehabil. 2019 Jul;26(5):399-404. doi: 10.1080/10749357.2019.1607485. Epub 2019 Apr 30. PMID 31038012
- [Result] LeLaurin JH, Lamba AH, Eliazar-Macke ND, Schmitzberger MK, Freytes IM, Dang S, Vogel WB, Levy CE, Klanchar SA, Beyth RJ, Shorr RI, Uphold CR. Postdischarge Intervention for Stroke Caregivers: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Nov 11;9(11):e21799. doi: 10.2196/21799. PMID 33174856

RESULTS

PARTICIPANT FLOW:
Period: Post-Test 1
Arm/Group | Caregiver Education and Support | Standard Care
Started | 86 | 88
Completed | 43 | 73
Not Completed | 43 | 15
Period: Post-Test 2
Arm/Group | Caregiver Education and Support | Standard Care
Started | 43 | 73
Completed | 43 | 71
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caregiver Education and Support | Standard Care | Total
Number analyzed (Participants) | 86 | 88 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (10.1) | 58.6 (13.7) | 59.1 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 80 | 154
  Male | 12 | 8 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 13 | 21
  Not Hispanic or Latino | 78 | 75 | 153
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 18 | 45
  White | 52 | 59 | 111
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 8 | 15
Education [Count of Participants; unit: Participants]
  ≤ High school | 27 | 20 | 47
  Some college/vocational school | 36 | 38 | 74
  College graduate | 23 | 30 | 53
Relationship to stroke survivor [Count of Participants; unit: Participants]
  Spouse/partner | 59 | 61 | 120
  Child | 9 | 16 | 25
  Other | 18 | 11 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change in Depressive Symptoms at 11 Weeks
Description: Changes in depressive symptoms will be measured with the Center for Epidemiologic Studies Depression (CES-D) scale. The CES-D is a 20-item, 4-point Likert scale ranging from never (0) to most of the time (3). Possible scores range from 0-60 with higher scores indicating more symptoms. It has been used in numerous studies with caregivers and has good reliability and validity.
Time Frame: 11 weeks after baseline
Population: All data collected from the 174 participants irrespective of their completion of the study were used in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | -1.8 (9.4) | -1.6 (9.0)
Statistical Analysis 1: Comparison: Caregiver Education and Support vs Standard Care; Test type: Superiority; p = 0.693, Mixed Models Analysis — a priori <.05 threshold; Slope = -0.68, Standard Error of Mean 1.72 — group X time interaction

2. Primary Outcome: Change in Depressive Symptoms at 19 Weeks
Description: as for outcome 1
Time Frame: 19 weeks after baseline
Population: All data collected from the 174 participants irrespective of their completion of the study were used in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | -1.3 (11.4) | 0.2 (11.0)
Statistical Analysis 1: Comparison: Caregiver Education and Support vs Standard Care; Test type: Superiority; p = 0.693, Mixed Models Analysis — a priori <.05 threshold; Slope = -2.17, Standard Error of Mean 2.07 — group x time interaction

3. Primary Outcome: Change in Caregiver Burden - Zarit
Description: Changes in burden will be measured by the Short Version of the Zarit Burden Interview (S-ZBI). This 12-item instrument was reduced from the original 29-item instrument. This instrument is scored on a 5-point Likert scale ranging from 0 (never) to 4 (nearly always). Possible scores range from 0-48 with higher scores indicating higher burden. The instrument was originally developed to measure dementia caregiver burden, but, the S-ZBI has been used in stroke caregiver studies and items are appropriate for other caregiver populations.
Time Frame: 11 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | -0.7 (5.7) | 1.3 (5.7)
Statistical Analysis 1: Comparison: Caregiver Education and Support vs Standard Care; Test type: Superiority; p = 0.055, Mixed Models Analysis; Slope = -2.08, Standard Error of Mean 1.08 — group X time interaction

4. Primary Outcome: Change in Caregiver Burden - Zarit
Description: as for outcome 3
Time Frame: 19 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | -0.6 (6.7) | 0.3 (5.6)
Statistical Analysis 1: Comparison: Caregiver Education and Support vs Standard Care; Test type: Superiority; p = 0.346, Mixed Models Analysis; Slope = -1.08, Standard Error of Mean 1.15 — group X time interaction

5. Primary Outcome: Change in Caregiver Burden - Time Required
Description: Changes in caregiver burden - time required will be measured by the Oberst Caregiving Burden Scale (OCBS). It contains 15 items that rate different types of caregiving tasks for stroke survivors based on perceived time and difficulty of the task. Each item is scored on a scale of 1 to 5 (total range from 15 to 75) with higher scores indicating greater time required or higher task difficulty.
Time Frame: 11 weeks after baseline
Population: All data collected from the 174 participants irrespective of their completion of the study were used in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | -16.8 (14.4) | -14.7 (12.9)

6. Primary Outcome: Change in Caregiver Burden - Time Required
Description: as for outcome 5
Time Frame: 19 weeks after baseline
Population: All data collected from the 174 participants irrespective of their completion of the study were used in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | -17.3 (12.7) | -14.5 (13.7)
Statistical Analysis 1: Comparison: Caregiver Education and Support vs Standard Care; Test type: Superiority; p = 0.688, Mixed Models Analysis — a priori <0.05; Slope = -0.72, Standard Error of Mean 1.79 — group X time interaction

7. Primary Outcome: Change in Caregiver Burden - Task Difficulty
Description: Changes in caregiver burden - task difficulty will be measured by the Oberst Caregiving Burden Scale (OCBS). The OCBS contains 15 items that rate different types of caregiving tasks for stroke survivors based on perceived time and difficulty of the task. Each item is scored on a scale of 1 to 5 (total range from 15 to 75) with higher scores indicating greater time required or higher task difficulty.
Time Frame: 11 weeks after baseline
Population: All data collected from the 174 participants irrespective of their completion of the study were used in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | -2.0 (8.4) | -0.5 (8.2)
Statistical Analysis 1: Comparison: Caregiver Education and Support vs Standard Care; Test type: Superiority; p = 0.418, Mixed Models Analysis — a priori <.05; Slope = -1.52, Standard Error of Mean 1.87 — group X time interaction

8. Primary Outcome: Change in Caregiver Burden - Task Difficulty
Description: as for outcome 7
Time Frame: 19 weeks after baseline
Population: All data collected from the 174 participants irrespective of their completion of the study were used in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | -2.5 (7.7) | -0.6 (8.3)
Statistical Analysis 1: Comparison: Caregiver Education and Support vs Standard Care; Test type: Superiority; p = 0.180, Mixed Models Analysis — a priori <0.05; Slope = -1.94, Standard Error of Mean 1.45 — group X time interaction

9. Secondary Outcome: Change in Perceived Stress
Description: Changes in perceived stress will be measured by the Perceived Stress Scale (PSS-4). The 4-item measure asses stress experienced in the last month on a 5-point Likert scale ranging from 0 (never) to 4 (very often). Scores range from 0-16, with higher scores indicating more stress.
Time Frame: 11 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | -0.5 (3.4) | -0.2 (3.0)
Statistical Analysis 1: Comparison: Caregiver Education and Support vs Standard Care; Test type: Superiority; p = 0.332, Mixed Models Analysis; Slope = -0.63, Standard Error of Mean 0.65 — group X time interaction

10. Secondary Outcome: Change in Perceived Stress
Description: as for outcome 9
Time Frame: 19 weeks after baseline
Population: All data collected from the 174 participants irrespective of their completion of the study were used in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | -0.6 (3.0) | -0.02 (3.2)
Statistical Analysis 1: Comparison: Caregiver Education and Support vs Standard Care; Test type: Superiority; p = 0.318, Mixed Models Analysis — a priori <0.05; Slope = -0.56, Standard Error of Mean 0.56 — group X time interaction

11. Secondary Outcome: Change in Positive Perceptions of Caregiving
Description: Changes in positive perceptions of caregiving will be measured by the Positive Aspects of Caregiving Scale. The scale contains 11 items scored from 1 (disagree a lot) to 5 (agree a lot). Total range from 11 to 55. Higher scores indicate more positive perceptions of caregiving.
Time Frame: 11 weeks after baseline
Population: All data collected from the 174 participants irrespective of their completion of the study were used in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | 2.1 (7.2) | 0.1 (6.7)
Statistical Analysis 1: Comparison: Caregiver Education and Support vs Standard Care; Test type: Superiority; p = 0.077, Mixed Models Analysis — a priori <.05; Slope = 2.33, Standard Error of Mean 1.31 — group X time interaction

12. Secondary Outcome: Change in Positive Perceptions of Caregiving
Description: as for outcome 11
Time Frame: 19 weeks after baseline
Population: All data collected from the 174 participants irrespective of their completion of the study were used in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | 1.1 (8.4) | 0.0 (7.2)
Statistical Analysis 1: Comparison: Caregiver Education and Support vs Standard Care; Test type: Superiority; p = 0.305, Mixed Models Analysis — a priori <0.05; Slope = 1.50, Standard Error of Mean 1.46 — group X time interaction

13. Secondary Outcome: Change in Stroke Knowledge
Description: Change in stroke knowledge will be measured by the Stroke Knowledge Instrument developed by the National Institutes of Health. This 7-item tool consists of true/false and multiple choice responses. Scores range from 0-7, with higher scores indicating more stroke knowledge.
Time Frame: 11 weeks after baseline
Population: All data collected from the 174 participants irrespective of their completion of the study were used in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | 1.3 (14.2) | 0.4 (15.8)

14. Secondary Outcome: Change in Stroke Knowledge
Description: as for outcome 13
Time Frame: 19 weeks after baseline
Population: All data collected from the 174 participants irrespective of their completion of the study were used in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | 0.0 (15.0) | 0.2 (15.0)

15. Secondary Outcome: Change in General Patient Satisfaction
Description: Changes in patient satisfaction will be measured by the General Satisfaction Subscale of the Long-Form Patient Satisfaction Questionnaire. This 6-item measure is scored from 1 (strongly agree) to 5 (strongly disagree). Total range from 6 to 30. Higher scores reflect better satisfaction with healthcare.
Time Frame: 11 weeks after baseline
Population: All data collected from the 174 participants irrespective of their completion of the study were used in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | -0.6 (5.5) | 0.1 (5.0)
Statistical Analysis 1: Comparison: Caregiver Education and Support vs Standard Care; Test type: Superiority; p = 0.514, Mixed Models Analysis — a priori <0.05; Slope = -0.62, Standard Error of Mean 0.94 — group X time interaction

16. Secondary Outcome: Change in General Patient Satisfaction
Description: as for outcome 15
Time Frame: 19 weeks after baseline
Population: All data collected from the 174 participants irrespective of their completion of the study were used in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | -1.6 (5.4) | 0.1 (5.1)
Statistical Analysis 1: Comparison: Caregiver Education and Support vs Standard Care; Test type: Superiority; p = 0.090, Mixed Models Analysis — a priori <0.05; Slope = -1.61, Standard Error of Mean 0.94 — group X time interaction

17. Secondary Outcome: Change in Veteran Functional Status
Description: Change in Veteran functional abilities will be measured by the Barthel Index, which measures patients' abilities to perform 10 self-care tasks. Response options vary for each item and are scored on 5-point increments (e.g., 0=unable, 5=needs help, 10-independent). Total scores range from 0-100 with higher scores indicating greater functional abilities.
Time Frame: 11 weeks after baseline
Population: All data collected from the 174 participants irrespective of their completion of the study were used in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | 8.5 (13.6) | 2.1 (13.3)
Statistical Analysis 1: Comparison: Caregiver Education and Support vs Standard Care; Test type: Superiority; p = 0.009, Mixed Models Analysis — a priori <0.05; Slope = 6.71, Standard Error of Mean 2.57 — group X time interaction

18. Secondary Outcome: Change in Veteran Functional Status
Description: as for outcome 17
Time Frame: 19 weeks after baseline
Population: All data collected from the 174 participants irrespective of their completion of the study were used in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | 5.6 (20.6) | 1.7 (17.2)
Statistical Analysis 1: Comparison: Caregiver Education and Support vs Standard Care; Test type: Superiority; p = 0.225, Mixed Models Analysis; Slope = 4.29, Standard Error of Mean 3.53 — group X time interaction

19. Secondary Outcome: Change in Self-efficacy - Obtaining Respite
Description: Measured by Revised Scale for Caregiver Self Efficacy - Obtaining Respite subscale (Steffen et al 2002). The subscale contains 5 items which ask caregivers to rate their level of confidence (from 0% to 100%) to ask for assistance. The subscale score is obtained by calculating the mean of the items, with a total score range of 0-100. Higher scores indicate higher self-efficacy. The subscale shows strong internal consistency and adequate test-retest reliability.
Time Frame: 11 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | 2.0 (23.7) | -1.1 (27.8)
Statistical Analysis 1: Comparison: Caregiver Education and Support vs Standard Care; Test type: Superiority; p = 0.443, Mixed Models Analysis — a priori <.05 threshold; Slope = 3.75, Standard Error of Mean 4.89 — group X time interaction

20. Secondary Outcome: Change in Self-efficacy - Obtaining Respite
Description: Measured by Revised Scale for Caregiver Self Efficacy - Obtaining Respite subscale (Steffen et al 2002). The subscale measures caregivers' confidence to ask for assistance. The subscale contains 5 items which ask caregivers to rate their level of confidence (from 0% to 100%) that they could perform the activity. The subscale score is obtained by calculating the mean of the items, with a total score range of 0-100. Higher scores indicate higher self-efficacy. The subscale shows strong internal consistency and adequate test-retest reliability.
Time Frame: 19 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | 4.5 (20.7) | -2.7 (31.96)
Statistical Analysis 1: Comparison: Caregiver Education and Support vs Standard Care; Test type: Superiority; p = 0.158, Mixed Models Analysis; Slope = 7.39, Standard Error of Mean 5.23 — group x time interaction

21. Secondary Outcome: Change in Self-efficacy - Controlling Upsetting Thoughts
Description: Measured by Revised Scale for Caregiver Self Efficacy - Controlling Upsetting Thoughts subscale (Steffen et al 2002). The subscale contains 5 items which ask caregivers to rate their level of confidence (from 0% to 100%) in their ability to control negative thoughts related to caregiving. The subscale score is obtained by calculating the mean of the items, with a total score range of 0-100. Higher scores indicate higher self-efficacy. The subscale shows strong internal consistency and adequate test-retest reliability.
Time Frame: 11 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | 4.7 (20.4) | -3.1 (18.3)
Statistical Analysis 1: Comparison: Caregiver Education and Support vs Standard Care; Test type: Superiority; p = 0.046, Mixed Models Analysis — a priori <.05 threshold; Slope = 7.28, Standard Error of Mean 3.64 — group X time interaction

22. Secondary Outcome: Change in Self-efficacy - Controlling Upsetting Thoughts
Description: as for outcome 21
Time Frame: 19 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | 4.5 (26.0) | -1.2 (18.4)
Statistical Analysis 1: Comparison: Caregiver Education and Support vs Standard Care; Test type: Superiority; p = 0.149, Mixed Models Analysis; Slope = 5.54, Standard Error of Mean 3.83 — group X time interaction

23. Secondary Outcome: Change in Health-Related Quality of Life - Physical
Description: Changes in health-related quality of life will be measured by the Rand 12-item Health Survey (VR-12). The VR12 items are scored on a 3-point or 5-point Likert scale. It consists of physical and emotional scales. Scores for each scale are calculated by using an algorithm and scores are standardized using a T-score metric with a mean of 50 and standard deviation of 10. Higher scores indicate better health-related quality of life. There is no composite or overall score for the VR-12.
Time Frame: 11 weeks after baseline
Population: All data collected from the 174 participants irrespective of their completion of the study were used in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | 2.2 (7.9) | -1.0 (8.5)
Statistical Analysis 1: Comparison: Caregiver Education and Support vs Standard Care; Test type: Superiority; p = 0.034, Mixed Models Analysis — a priori <0.05; Slope = 4.16, Standard Error of Mean 1.95 — group X time interaction

24. Secondary Outcome: Change in Health-Related Quality of Life - Physical
Description: as for outcome 23
Time Frame: 19 weeks after baseline
Population: All data collected from the 174 participants irrespective of their completion of the study were used in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | -1.2 (7.4) | -0.2 (8.5)
Statistical Analysis 1: Comparison: Caregiver Education and Support vs Standard Care; Test type: Superiority; p = 0.846, Mixed Models Analysis — a priori <0.05; Slope = -0.30, Standard Error of Mean 1.52 — group X time interaction

25. Secondary Outcome: Change in Health-Related Quality of Life - Mental Health
Description: as for outcome 23
Time Frame: 11 weeks after baseline
Population: All data collected from the 174 participants irrespective of their completion of the study were used in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | 1.4 (7.9) | 0.6 (9.1)
Statistical Analysis 1: Comparison: Caregiver Education and Support vs Standard Care; Test type: Superiority; p = .0442, Mixed Models Analysis — a priori <0.05; Slope = 1.67, Standard Error of Mean 2.17 — group X time interaction

26. Secondary Outcome: Change in Health-Related Quality of Life - Mental Health
Description: as for outcome 23
Time Frame: 19 weeks after baseline
Population: All data collected from the 174 participants irrespective of their completion of the study were used in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Education and Support | Standard Care
Number analyzed (Participants) | 86 | 88
score on a scale | 2.0 (9.5) | 0.6 (10.9)
Statistical Analysis 1: Comparison: Caregiver Education and Support vs Standard Care; Test type: Superiority; p = 0.293, Mixed Models Analysis — a priori <0.05; Slope = 1.98, Standard Error of Mean 1.88 — group X time interaction

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during participation in study (19 weeks).
Description: Caregivers were asked about adverse events during data collection sessions at 11 and 19 weeks.
Arm/Group | Caregiver Education and Support | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/88
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/88
Other Adverse Events (participants affected / at risk) | 0/86 | 1/88
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caregiver Education and Support (N=86) | Standard Care (N=88)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The intervention effects must be interpreted with caution. The study had reduced statistical power, which may have reduced the chances of detecting true effects of the intervention on some of the outcomes. Based on our original power analysis, we planned for a sample size of 240, but enrolled only 174 caregivers. Also, the effect size of the intervention may be overestimated as the intervention group had a higher attrition rate than the usual care group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-19): https://cdn.clinicaltrials.gov/large-docs/31/NCT01600131/Prot_SAP_000.pdf